CLINICAL TRIAL: NCT01434472
Title: A Phase II Trial of High-Dose 90Y-Ibritumomab Tiuxetan (Anti-CD20) Followed by Fludarabine and Low-Dose Total Body Irradiation and HLA-Matched Allogeneic Hematopoietic Transplantation for Patients With Relapsed or Refractory Aggressive B-Cell Lymphoma
Brief Title: High-Dose Y-90-Ibritumomab Tiuxetan Added to Reduced-Intensity Allogeneic Stem Cell Transplant Regimen for Relapsed or Refractory Aggressive B-Cell Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to insufficient funding
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ajay Gopal, Professor, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2398.00; NCI-2011-01189 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2398.00 (Other: Fred Hutch/University of Washington Cancer Consortium); P01CA044991 (NIH); P30CA015704 (NIH); RG9213033 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2011-07-26; First posted 2011-09-15 (Estimated); Results first posted 2021-05-25 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Post-Transplant Lymphoproliferative Disorder; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent B-Cell Non-Hodgkin Lymphoma; Recurrent Burkitt Lymphoma; Refractory B-Cell Non-Hodgkin Lymphoma; Refractory Burkitt Lymphoma; Refractory Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, B-Cell; Burkitt Lymphoma | interventions — Cyclosporine; Cyclosporins; fludarabine phosphate; Indium; Mycophenolic Acid; Rituximab; CT-P10; Whole-Body Irradiation; ibritumomab tiuxetan; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (radiolabeled antibody, TBI, allogeneic PBSCT) (Experimental): Beginning 24-48 hours prior to therapy infusion, patients receive rituximab IV over 4-6 hours and then receive a therapy-dose of high-dose yttrium Y 90 ibritumomab tiuxetan IV over 30 minutes on day -14 prior to transplant. Patients also receive fludarabine phosphate IV on days -4 to -2 and undergo TBI followed by allogeneic PBSCT on day 0. Patients also receive cyclosporine PO BID on days -3 to 56 with taper to day 180 (related donor) or -3 to 100 with taper over 11 weeks (unrelated donor) and mycophenolate mofetil PO BID on days 0-27 (related donor) or PO TID on days 0-40 with taper to day 96 (unrelated donor).
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Cyclosporine; Drug: Fludarabine Phosphate; Radiation: Indium In-111 Ibritumomab Tiuxetan; Drug: Mycophenolate Mofetil; Other: Pharmacological Study; Biological: Rituximab; Radiation: Total-Body Irradiation; Radiation: Yttrium Y-90 Ibritumomab Tiuxetan; Drug: Fludarabine

INTERVENTIONS:
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo allogeneic PBSCT (infusion of donor stem cells via central catheter)
  Other Names: allogeneic stem cell transplantation; HSC; HSCT
Drug: Cyclosporine — Given PO
  Other Names: 27-400; Ciclosporin; CsA; Cyclosporin; Cyclosporin A; Gengraf; Neoral; OL 27-400; Sandimmun; Sandimmune; SangCya
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586
Radiation: Indium In-111 Ibritumomab Tiuxetan — Given IV
  Other Names: IDEC In2B8; IDEC-In2B8; In 111 Ibritumomab Tiuxetan; In 111 Zevalin; indium In 111 ibritumomab tiuxetan
Drug: Mycophenolate Mofetil — Given PO
  Other Names: Cellcept; MMF
Other: Pharmacological Study — Correlative studies
Biological: Rituximab — Given IV prior to yttrium Y 90 ibritumomab tiuxetan
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; RTXM83
Radiation: Total-Body Irradiation — Undergo TBI
  Other Names: TOTAL BODY IRRADIATION; Whole-Body Irradiation; TBI; Whole Body Irradiation
Radiation: Yttrium Y-90 Ibritumomab Tiuxetan — Given IV
  Other Names: IDEC-Y2B8; IDEC-Y2B8 monoclonal antibody; Y 90 Ibritumomab Tiuxetan; Y 90 Zevalin; Yttrium Y 90 Ibritumomab Tiuxetan; yttrium Y90 ibritumomab tiuxetan
Drug: Fludarabine — Given IV
  Other Names: 118218; 2-Fluoro-9-beta-arabinofuranosyladenine; 2-Fluorovidarabine; 9-Beta-D-arabinofuranosyl-2-fluoro-9H-purin-6-amine; Fluradosa

SUMMARY:
This phase II trial studies the side effects and how well high-dose yttrium-90 (Y-90)-ibritumomab tiuxetan (anti-cluster of differentiation [CD]20) followed by fludarabine phosphate, low-dose total body irradiation (TBI), and donor peripheral blood stem cell transplant (PBSCT) work in treating patients with aggressive B-cell lymphoma that has returned after a period of improvement (relapsed) or has not responded to previous treatment (refractory). Radiolabeled monoclonal antibodies, such as Y-90-ibritumomab tiuxetan, can find cancer cells and carry cancer-killing substances to them with less effect on normal cells. Giving chemotherapy, such as fludarabine phosphate, and TBI before a donor PBSCT helps stop the growth of cancer cells. It may also stop the patient's immune system from rejecting the donor's stem cells. However, high-dose radiolabeled antibodies also destroy healthy blood cells in the patient's body. When healthy stem cells from a donor are infused into the patient (stem cell transplant), they may help the patient's body replace these blood cells. Giving high-dose Y-90-ibritumomab tiuxetan followed by fludarabine phosphate, TBI, and donor PBSCT may be an effective treatment for patients with B-cell lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety and efficacy of 1.5 mCi/kg (max 120 mCi) 90Y-Ibritumomab tiuxetan (yttrium Y 90 ibritumomab tiuxetan) (anti-CD20) combined with fludarabine (fludarabine phosphate) (30 mg/m^2 x 3) and 2 gray (Gy) total body irradiation followed by human leukocyte antigens (HLA) matched allogeneic hematopoietic transplantation for patients with relapsed or refractory aggressive B-cell lymphoma.

OUTLINE:

Beginning 24-48 hours prior to therapy infusion, patients receive rituximab intravenously (IV) over 4-6 hours and then receive a therapy-dose of high-dose yttrium Y 90 ibritumomab tiuxetan IV over 30 minutes on day -14 prior to transplant. Patients also receive fludarabine phosphate IV on days -4 to -2 and undergo TBI followed by allogeneic PBSCT on day 0. Patients also receive cyclosporine orally (PO) twice daily (BID) on days -3 to 56 with taper to day 180 (related donor) or -3 to 100 with taper over 11 weeks (unrelated donor) and mycophenolate mofetil PO BID on days 0-27 (related donor) or PO thrice daily (TID) on days 0-40 with taper to day 96 (unrelated donor).

After completion of study treatment and assessments through ~day 100 following transplant, patients are followed up at 1, 3, 6, and 12 months and then annually up to 2 years thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically confirmed diagnosis of aggressive B-cell lymphoma (diffuse large B-cell lymphoma [DLBCL], Burkitt lymphoma [BL], etc.) expressing the CD20 antigen and have failed at least one prior standard systemic therapy
* Patients must have relapsed after high-dose therapy and autologous transplantation or be ineligible for high-dose therapy and autologous transplantation; patients that have failed autologous transplantation are those with persistent disease > 30 days after transplant; those ineligible for autologous transplant include those with chemoresistant disease (i.e., patients who have not achieved a partial response or better with their most recent chemotherapy regimen), are expected to have a poor outcome from autologous transplant (e.g., DLBCL relapsing within one year of rituximab, cyclophosphamide, doxorubicin hydrochloride, vincristine sulfate, prednisone [R-CHOP]-like chemotherapy, double hit lymphoma, v-myc myelocytomatosis viral oncogene homolog (avian) positive [MYC+] lymphoma, persistent positron emission tomography [PET] positivity after chemotherapy), are unable to collect sufficient or tumor-free autologous stem cells per Seattle Cancer Care Alliance (SCCA) standard practice, are unable to tolerate the high-dose autologous conditioning regimens, or who refuse a high-dose autologous transplant regimen
* Creatinine (Cr) < 2.0
* Bilirubin < 1.5 mg/dL with the exception of patients thought to have Gilbert's syndrome, who may have a total bilirubin above 1.5 mg/dL
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) < 3 x upper limit of normal (ULN)
* Patients must have an expected survival without treatment of > 60 days and must be free of major infection including human immunodeficiency virus (HIV)
* Patients must have an HLA-identical related or HLA-matched unrelated donor

Exclusion Criteria:

* Receipt of systemic anti-lymphoma therapy withinthe following intervals prior to the therapeutic 90Y-ibritumomab tiuxetan dose:

  * < 30 days for intravenously-administered cytotoxic chemotherapy and/or monoclonal antibodies
  * < 5 half-lives for all other anti-cancer agents (e.g., targeted therapies, corticosteroids, immunomodulatory agents, etc.)
* Inability to understand or give an informed consent
* Active central nervous system lymphoma
* Pregnancy
* Fertile men or women unwilling to use contraceptive techniques during and for 12 months following treatment
* Southwest Oncology Group (SWOG)/Eastern Cooperative Oncology Group (ECOG) performance score >= 2
* High-dose chemotherapy or external beam radiation therapy to lung, liver, or kidneys > 20 Gy within the previous 100 days prior to therapeutic 90Y-ibritumomab tiuxetan dose
* Medical condition that would contraindicate allogeneic transplantation as per standard practice guidelines (e.g., impaired cardiopulmonary function, hepatitis, etc)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-11-16 (Actual); Primary Completion 2020-05-06 (Actual); Study Completion 2020-05-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Gopal, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Radiolabeled Antibody, TBI, Allogeneic PBSCT)
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Radiolabeled Antibody, TBI, Allogeneic PBSCT)
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 1
Age, Continuous [Median (Full Range); unit: years] | 52.5 [36 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Based on a one-sample chi-square test with one-sided significance level of five percent. This study will be deemed successful if the 1 year progression-free survival of this highest-risk group of patients is 54% or greater.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Radiolabeled Antibody, TBI, Allogeneic PBSCT)
Number analyzed (Participants) | 20
Participants | 11

2. Secondary Outcome: Absolute Neutrophil Count (ANC) Engraftment
Description: The median time in days to achieve ANC recovery defined as ANC>500uL.
Time Frame: Up to day 100
Measure: Median (Full Range); unit: Days
Arm/Group | Treatment (Radiolabeled Antibody, TBI, Allogeneic PBSCT)
Number analyzed (Participants) | 20
Days | 16 [7 to 24]

3. Secondary Outcome: Overall Survival
Time Frame: Up to 2 years post transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Radiolabeled Antibody, TBI, Allogeneic PBSCT)
Number analyzed (Participants) | 20
Participants | 14

4. Secondary Outcome: Response Rates
Description: Response is defined as having achieved a Partial Response or better.
Time Frame: Day 100
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Radiolabeled Antibody, TBI, Allogeneic PBSCT)
Number analyzed (Participants) | 20
Participants | 16

5. Secondary Outcome: Treatment-related Mortality
Description: Defined as death in the absence of progressive lymphoma that can be possibly, probably, or definitely attributed to the radioimmunotherapy.
Time Frame: Day 100
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Radiolabeled Antibody, TBI, Allogeneic PBSCT)
Number analyzed (Participants) | 20
Participants | 1

6. Secondary Outcome: Platelet Engraftment
Description: The median time in days to achieve platelet recovery as defined as platelet >20,000uL.
Time Frame: Up to day 100
Measure: Median (Full Range); unit: Days
Arm/Group | Treatment (Radiolabeled Antibody, TBI, Allogeneic PBSCT)
Number analyzed (Participants) | 20
Days | 9 [0 to 21]

7. Secondary Outcome: Hematopoietic Toxicity
Description: Clinical sequelae due to hematopoietic toxicity as defined by incidences of neutropenic fever and bleeding.
Time Frame: Up to day 100
Measure: Number; unit: Incidences
Arm/Group | Treatment (Radiolabeled Antibody, TBI, Allogeneic PBSCT)
Number analyzed (Participants) | 20
Incidences | 5

ADVERSE EVENTS:
Time Frame: AEs will be collected from the time of first exposure to a study intervention (i.e., the start of the rituximab infusion associated with the therapy dose) through day +100 post-transplant or through discharge prior to that date from the SCCA system to care of the patient's primary physician.
Arm/Group | Treatment (Radiolabeled Antibody, TBI, Allogeneic PBSCT)
All-Cause Mortality (participants affected / at risk) | 6/20
Serious Adverse Events (participants affected / at risk) | 11/20
Other Adverse Events (participants affected / at risk) | 11/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Radiolabeled Antibody, TBI, Allogeneic PBSCT) (N=20)
Thromboembolic event - cerebal infarct (Vascular disorders) | 1 (1)
Wound Infection (Infections and infestations) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 2 (2)
Acute Renal Injury (Investigations) | 2 (2)
Adenovirus pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
ARDS (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Ascites (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (3)
Dizziness (Nervous system disorders) | 1 (1)
E. coli bacteremia (Infections and infestations) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1)
Extrapyramidal disorder (Nervous system disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Blood infection (Infections and infestations) | 2 (2)
Neutropenic fever (Infections and infestations) | 3 (5)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Radiolabeled Antibody, TBI, Allogeneic PBSCT) (N=20)
Anorexia (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 3 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-07): https://cdn.clinicaltrials.gov/large-docs/72/NCT01434472/Prot_SAP_000.pdf